CLINICAL TRIAL: NCT04842396
Title: Low-volume Cycling Training Improves Body Composition and Functionality in Older People With Multimorbidity
Brief Title: Low-volume Cycling Training in Older People With Multimorbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Responsible Party: Principal Investigator, José Carlos Millán Calenti, Full Professor, Universidade da Coruña
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/010; ED431C 2017/49 (Other Grant/Funding Number: Xunta de Galicia); ED431F 2017/09 (Other Grant/Funding Number: Xunta de Galicia); IN607C 2016/08 (Other Grant/Funding Number: Xunta de Galicia); IN607C 2017/02 (Other Grant/Funding Number: Xunta de Galicia); RYC-2015-18394 (Other Grant/Funding Number: Spanish Ministry of Economy and Competitiveness)
Record Dates: First submitted 2021-04-06; First posted 2021-04-13 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Frailty; Morbidity, Multiple
Keywords: physical exercise; body composition; physical functionality; blood pressure; individualized training; morbidity
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Motorized cycle ergometer (Experimental): The exercise group cycles 20 minutes per session on the MOTOmed Muvi 3 days per week for 6 weeks at an intensity guided by the perception of effort.
  A cycling cadence is fixed between 25 and 30 rpm for all sessions since that cadence is comfortable for every participant. Researchers adjust resistance on the motorized cycle to increase the external load until it reached the level required to reach the intensity of effort programmed by the OMNI-RPE. The six weeks are programmed in the form of two intensity-differentiated training phases of three weeks. In the first training phase (i.e., the first three weeks), participants are requested to cycle simultaneously with the upper and lower limbs at an intensity equivalent to a perception of 3 (i.e., easy to somewhat moderate) on the OMNI-RPE (0-10).
  Interventions: Other: Experimental:Motorized cycle ergometer
- Control group (No Intervention): Participants are evaluated the week before and the week after the experimental group finishes the training period (pre- vs. postintervention) to facilitate an examination of the changes in body composition, functional performance, and resting cardiovascular state.

INTERVENTIONS:
Other: Experimental:Motorized cycle ergometer — Cycling training on the MOTOmed Muvi for 20 minutes 3 days per week for 6 weeks. Moreover, control of adverse events throughout the trial was measured through the assessment and monitoring of vital signs before, during (within the first 10 minutes), and after the intervention sessions. Vital signs [heart rate (per minute), systolic and diastolic blood pressure (in millimeters of mercury, mm Hg), and oxygen saturation (in percentage)] were monitored by a nurse and a medical doctor using mobile finger pulse oximeters.
  Arms: Experimental: Motorized cycle ergometer

SUMMARY:
INTRODUCTION: Physical exercise, when practiced regularly and in adequate doses, is a proven nonpharmacological measure that helps to prevent and reverse noncommunicable diseases, as well as reduce mortality rates from any cause. In general, older adults perform insufficient physical activity and do not meet the doses recommended by the World Health Organization for the improvement of health through physical activity.

OBJECTIVE: Our main aim will be to evaluate the effect of a 6-week intervention on health-related outcomes (body composition, hemodynamic and functionality changes) in 24 individuals aged 65 and older with multimorbidity.

METHODS AND ANALYSIS: The study was a 2 x 2 randomized controlled trial using a two-group design (exercise vs. control) and two repeated measures (pre- vs. postintervention). The intervention (on the MOTOmed Muvi) will consist of a very low volume (60 minutes per week) of low-to-moderate intensity exercise training to assess body composition evaluation, hemodynamic parameter evaluation and functional evaluation. Participants will be recruited at the Gerontological Complex La Milagrosa (A Coruña, Spain), consisting of a daycare center and a nursing home.

For the statistical analysis, nonparametric ANOVA type statistics and mixed models for repeated measures will be used.

DETAILED DESCRIPTION:
INTRODUCTION. Aging is a risk factor for most chronic diseases, and the presence of more than two diseases (i.e., multimorbidity), which is frequent in almost two out of three older adults, has been related to an increased risk of disability and frailty, a decrease in quality of life, and mortality. Physical activity (PA) acts as a nonpharmacological intervention and regular physical activity (rPA) reduces rates of all-cause mortality, compresses morbidity, decreases healthcare costs, and has relatively minimal adverse effects compared to drugs. It has been estimated that 27.5% of the world's population in 2016 did not meet the recommendations established for the member states of the World Health Organization (WHO) for health-enhancing physical activity. Furthermore, recent studies showed that moderate-intensity physical activity may be sufficient for reducing the risk of all-cause dementia and that some of the protective benefits of physical activity for older adults. It seems indispensable to study adequate doses of exercise for older people who often have low levels of physical activity and fitness, who spend a large amount of time sitting down, and whose multimorbidity keeps them away from exercising.

OBJECTIVE: To study the effects of perception-regulated low-volume and low-to-moderate intensity training on body composition, hemodynamic parameters, and functional performance in older adults with multimorbidity.

MATERIAL AND METHODS: The study is a 2 x 2 randomized controlled trial using a two-group design (exercise vs. control) and two repeated measures (pre- vs. postintervention). The exercise group is requested to accomplish on the MOTOmed Muvi, a low volume (i.e., 20 minutes, 3 days per week) and low-to-moderate intensity combining upper and lower limb recumbent cycling training for six weeks. Participants are evaluated to examine the changes in body composition, functional performance, and resting cardiovascular state. Furthermore, participants are monitored physiologically during each session (HR and blood pressure) to control any possible adverse effects. Participants are recruited at the Gerontological Complex La Milagrosa (A Coruña, Spain), consisting of a daycare center and a nursing home. 24 participants will be recruited and randomly placed into two groups: the exercise group (EG, n=12) and the control group (CG, n=12). A stratified permuted block randomization is employed that accounted for the GDS score, sex, and type of institutionalization.

DATA ANALYSIS AND STATISTICS: Data will be presented as the median and interquartile range for ordinal variables and the estimated marginal mean ± standard deviation (SD) for continuous variables. The effect of the intervention will be analyzed employing nparLD (nonparametric analysis of longitudinal data in factorial experiments) from the R software package. Changes within and between groups will be analyzed by employing mixed models for repeated measures designs with the module GAMLj, which uses the R formulation of random effects as implemented by the lme4 R package in Jamovi software.

ELIGIBILITY:
Inclusion criteria:

* men and women aged 65 and older
* users of a care setting-daycare patients or nursing home residents
* a score < 5 in the Global Deterioration Scale (GDS), from no cognitive decline to moderate cognitive decline.

Exclusion criteria:

* physical limitations or musculoskeletal injuries that could affect cycling training performance; physical exercise contraindicated by the physiotherapist and verified by the medical doctor according to the medical register of each participant
* heart failure with a functional class according to the New York Heart Association (NYHA) Classification of NYHA III and IV
* the presence of acute pain that does not allow exercise training
* recent acute myocardial infarction (in last 6 months) or unstable angina
* uncontrolled hypotension
* uncontrolled arterial hypertension (>180/100 mmHg)
* active cancer treatment with chemotherapy
* patients with an active pacemaker and/or uncontrolled block
* diabetes mellitus with acute decompensation or uncontrolled hypoglycemia
* any other circumstance that precludes individuals from completing the training intervention.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Body weight | 6 weeks
  Body composition evaluation by Bioimpedance analysis (Inbody 270): body weight (in kg)
Muscle mass | 6 weeks
  Body composition evaluation by bioimpedance analysis (Inbody 270): muscle mass (MM, in kg)
Fat mass | 6 week
  Body composition evaluation by bioimpedance analysis (Inbody 270): fat mass (FM, in kg).
Fat mass percentage | 6 week
  Body composition evaluation by bioimpedance analysis (Inbody 270): fat mass percentage.
Waist circumference | 6 weeks
  Waist circumference (WC, cm) is taken at end tidal using a measuring tape to the nearest 0.1 cm, midway between the lowest rib and the iliac crest, which corresponded with the level of the umbilicus.
Heart rate | 6 weeks
  The baseline hemodynamic state is characterized by storing the mean of the three lowest values for thirty seconds of heart rate (HRrest; in BPM, beats per minute) with a finger pulse oximeter.
Systolic blood pressure | 6 weeks
  Blood pressure (mm Hg) by the auscultator method using a properly calibrated mercury column sphygmomanometer flexible cuff of the appropriate size and a stethoscope. Three systolic (SBPrest) measurements are recorded at 1-minute intervals.
Diastolic blood pressure | 6 weeks
  Blood pressure (mm Hg) by the auscultator method using a properly calibrated mercury column sphygmomanometer flexible cuff of the appropriate size and a stethoscope.Three diastolic blood pressure (DBPrest) measurements are recorded at 1-minute intervals.
Mean blood pressure | 6 weeks
  Mean blood pressure (MBPrest, in mm Hg) is calculated as follows:
  MBP=DBP+1/3 (SBP-DBP)
The Performance-Oriented Mobility Assessment (POMA) | 6 weeks
  Functional evaluation: The Performance-Oriented Mobility Assessment (i.e., POMA), which measures balance (i.e., POMA-B; scored over 16) and gait performance (i.e., POMA-G; scored over 12) and the total score (i.e., POMA-T; scored over 28). A lower score implies a higher risk of falling. 25-28= low fall risk; 19-24= medium fall risk; and <19= high fall risk.
The Short Physical Performance Battery test (SPPB) | 6 weeks
  Functional evaluation: The Short Physical Performance Battery test (i.e., SPPB) to evaluate the time spent to complete three components:
  1. three balance tasks (i.e., SPPB-B): side-by-side stand, semi-tandem stand, and tandem stand
  2. gait speed test; walk 4 meters at a comfortable speed (i.e., SPPB-G)
  3. chair stand test; sit-to-stand 5 times from a chair (i.e., SPPB-ChS). Each component is scored out of 4, giving a maximum of 12 and a minimum of 0. A higher score implies better function and lower fall rate.
Chair Sit-and-Reach Test (CSR) | 6 weeks
  Functional evaluation: Chair Sit-and-Reach Test (CSR) to measure lower body flexibility. The score (in cm) is the most distant point reached with the fingertips. Lower distances implies lower flexibility.
Frailty | 6 weeks
  Functional evaluation: Frailty assessed by Fried et al. (2001) phenotype, consisting of five components: unintentional weight loss, self-reported exhaustion, weakness (grip strength), slow walking speed, and low physical activity. Individuals are classified as robust (zero positive components), pre-frail (one or two positive components) and frail (three or more positive components).

CONTACTS AND LOCATIONS:
Overall Officials: José C. Millán-Calenti, PhD, Principal Investigator — Universidade da Coruña
Locations (1):
- Universidade da Coruña, A Coruña, Spain

REFERENCES:
- [Background] Nunes BP, Flores TR, Mielke GI, Thume E, Facchini LA. Multimorbidity and mortality in older adults: A systematic review and meta-analysis. Arch Gerontol Geriatr. 2016 Nov-Dec;67:130-8. doi: 10.1016/j.archger.2016.07.008. Epub 2016 Aug 2. PMID 27500661
- [Background] Booth FW, Roberts CK, Laye MJ. Lack of exercise is a major cause of chronic diseases. Compr Physiol. 2012 Apr;2(2):1143-211. doi: 10.1002/cphy.c110025. PMID 23798298
- [Background] Pedersen BK. The Physiology of Optimizing Health with a Focus on Exercise as Medicine. Annu Rev Physiol. 2019 Feb 10;81:607-627. doi: 10.1146/annurev-physiol-020518-114339. Epub 2018 Dec 10. PMID 30526319
- [Background] Fiuza-Luces C, Garatachea N, Berger NA, Lucia A. Exercise is the real polypill. Physiology (Bethesda). 2013 Sep;28(5):330-58. doi: 10.1152/physiol.00019.2013. PMID 23997192
- [Background] Cunningham C, O' Sullivan R, Caserotti P, Tully MA. Consequences of physical inactivity in older adults: A systematic review of reviews and meta-analyses. Scand J Med Sci Sports. 2020 May;30(5):816-827. doi: 10.1111/sms.13616. Epub 2020 Feb 4. PMID 32020713
- [Background] Reisberg B, Ferris SH, de Leon MJ, Crook T. The Global Deterioration Scale for assessment of primary degenerative dementia. Am J Psychiatry. 1982 Sep;139(9):1136-9. doi: 10.1176/ajp.139.9.1136. PMID 7114305
- [Background] Tinetti ME. Performance-oriented assessment of mobility problems in elderly patients. J Am Geriatr Soc. 1986 Feb;34(2):119-26. doi: 10.1111/j.1532-5415.1986.tb05480.x. No abstract available. PMID 3944402
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Guidetti L, Sgadari A, Buzzachera CF, Broccatelli M, Utter AC, Goss FL, Baldari C. Validation of the OMNI-cycle scale of perceived exertion in the elderly. J Aging Phys Act. 2011 Jul;19(3):214-24. doi: 10.1123/japa.19.3.214. PMID 21727302
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Mezzani A, Hamm LF, Jones AM, McBride PE, Moholdt T, Stone JA, Urhausen A, Williams MA; European Association for Cardiovascular Prevention and Rehabilitation; American Association of Cardiovascular and Pulmonary Rehabilitation; Canadian Association of Cardiac Rehabilitation. Aerobic exercise intensity assessment and prescription in cardiac rehabilitation: a joint position statement of the European Association for Cardiovascular Prevention and Rehabilitation, the American Association of Cardiovascular and Pulmonary Rehabilitation and the Canadian Association of Cardiac Rehabilitation. Eur J Prev Cardiol. 2013 Jun;20(3):442-67. doi: 10.1177/2047487312460484. Epub 2012 Oct 26. PMID 23104970
- [Derived] Carballeira E, Censi KC, Maseda A, Lopez-Lopez R, Lorenzo-Lopez L, Millan-Calenti JC. Low-volume cycling training improves body composition and functionality in older people with multimorbidity: a randomized controlled trial. Sci Rep. 2021 Jun 28;11(1):13364. doi: 10.1038/s41598-021-92716-9. PMID 34183717
- See also: 9. World Health Organization. Global action plan on physical activity 2018-2030: more active people for a healthier world — https://apps.who.int/iris/bitstream/handle/10665/272722/9789241514187-eng.pdf?ua=1
- See also: 10. World Health Organization. Global recommendations on physical activity for health — https://apps.who.int/iris/bitstream/handle/10665/44399/9789241599979_eng.pdf?sequence=1.

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT04842396/SAP_001.pdf